CLINICAL TRIAL: NCT07301580
Title: Physical Prehabilitation of Breast Cancer-Related Lymphedema
Brief Title: Prehabilitation of Breast Cancer-Related Lymphedema
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Health Sciences Balikesir Hospital Eduation and Research (Other Government)
Responsible Party: Principal Investigator, Mustafa Akin, Associated Professor, University of Health Sciences Balikesir Hospital Eduation and Research
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: UHSBalikesirRadiationOnc
Record Dates: First submitted 2025-11-27; First posted 2025-12-24 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-10

CONDITIONS: Breast Cancer-Related Arm Lymphedema; Quality of Life Impairment; Fatigue Syndrome, Chronic; Prehabilitation
Keywords: Breast cancer-related lymphedema; prehabilitation; pre-irradiation; pre-surgery
MeSH Terms: conditions — Breast Cancer Lymphedema; Fatigue Syndrome, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Prehabilitation Exercise Group (Other): Behavioral Intervention
  Interventions: Behavioral: Prehabilitation Exercise Group

INTERVENTIONS:
Behavioral: Prehabilitation Exercise Group — A personalized upper-extremity exercise program initiated before surgery and continued for 12 months postoperatively. The program includes mobility, stretching, strengthening, and functional exercises tailored to individual needs. Instruction is provided through written and visual materials, with follow-up contacts to reinforce adherence.

SUMMARY:
This prospective prehabilitation study aims to evaluate the effects of an individualized exercise program initiated before breast cancer surgery and continued for 12 months postoperatively. The intervention focuses on incidence of breast cancer-related lymphedema, improving functional outcomes, range of motion, pain, and patient-reported measures throughout the surgical and recovery phases. Participants receive structured, personalized exercise instructions and are monitored regularly during follow-up.

The study assesses the trajectory of extremity volume difference, early postoperative pain, the recovery pattern of shoulder range of motion and changes in functional status across the first postoperative year. Additionally, it examines the incidence of lymphedema and explores demographic and clinical determinants affecting patient outcomes. The findings are expected to provide evidence for the integration of prehabilitation into standard breast cancer care pathways.

DETAILED DESCRIPTION:
This prospective prehabilitation study investigates the effectiveness of an individualized exercise program initiated before breast cancer surgery and radiation therapy maintained for 12 months postoperatively. The intervention was designed to optimize physical readiness for surgery, support early postoperative recovery, and promote long-term functional improvement. Participants received structured exercise instructions delivered through visual and written materials, and adherence was reinforced through regular follow-up contacts.

The primary focus of the study is to characterize postoperative functional trajectories, including pain intensity, shoulder range of motion (ROM), upper-extremity function, and patient-reported outcomes. Particular emphasis is placed on the early postoperative period, during which pain typically increases and functional limitations become more pronounced. Longitudinal assessments allow observation of recovery patterns across all ROM planes, with anticipated improvements in flexion and abduction by the third postoperative month and further recovery in internal and external rotation by the sixth month.

A secondary objective is to monitor the development of lymphedema, defined by limb volume differences and physical signs of edema. The study also explores demographic and clinical determinants that may influence treatment outcomes, aiming to identify subgroups that benefit most from prehabilitation. By evaluating functional, symptomatic, and quality-of-life outcomes across a 12-month period, this study provides evidence to support the incorporation of preoperative exercise interventions into standard breast cancer care pathways.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18 years or older
* Diagnosed with breast cancer and scheduled for surgical treatment
* Able to perform prescribed upper-extremity exercises
* Able to provide informed consent and complete follow-up assessments.

Exclusion Criteria:

* Presence of metastatic disease at baseline
* Neurological, orthopedic, or systemic conditions limiting upper-extremity mobility
* Prior breast or axillary surgery on the same side
* Planned neoadjuvant chemotherapy that would delay the initiation of the exercise program
* Inability to comply with the exercise instruction or follow-up schedule

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — female breast cancer survivors
Enrollment: 40 (Actual)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-10-05 (Actual); Study Completion 2025-10-05 (Actual)

PRIMARY OUTCOMES:
Incidence of Lymphedema Development | Baseline; 1, 3, 6, and 12 months postoperatively
  Lymphedema is determined by volume differences between extremities and physical signs of edema.
  Physical examination consists of inspection of the patient for swelling, rash, dermal ulcerations, hyperkeratosis, vascular signs continuing with palpation for pitting and Stemmer's sign. Limb circumferences were measured using a constant-tension tape beginning from the ulnar styloid process in the upper extremity with 4 cm intervals up to 32 cm. Afterwards limb volume was estimated via calculator model.
  Calculation results are compared by opposite limb and volume difference of 200 ml or 5-10% is considered as Lymphedema. Clinical severity was graded according to the International Society of Lymphology (ISL) staging system (Stages 0-III), based on presence of swelling, reversibility, pitting, and tissue fibrosis.
Pain Intensity | Baseline; 1, 3, 6, and 12 months postoperatively
  The Visual Analogue Scale (VAS) measures pain intensity. The VAS consists of a 10cm line, with two end points representing 0 ('no pain') and 10 ('pain as bad as it could possibly be'). It is performed by asking the patient to rate their current level of pain by placing a mark on the line.
Quality of Life Impairment | Baseline; 3, 6, and 12 months postoperatively
  Quality of life is assessed with standardized patient-reported questionnaires. The EORTC Core Quality of Life(QoL) questionnaire (EORTC QLQ-C30) is designed to measure cancer patients' physical, psychological and social functions. The questionnaire is composed of multi-item scales and single items.
  EORTC-QLQ-C30 gives information about how affected the patients are about physical, emotional, social and financial aspects because of the disease and treatments. Form includes twenty-eight questions answered as from one to four Likert scale, reflecting grades of agree to disagree respectively. Final two questions necessitate giving value on a seven point scale, to the quality of life and global health of the last week. Global health score and physical functioning score reflects better QoL in higher values while symptom scale results worser in high values.

SECONDARY OUTCOMES:
Upper Extremity Function | Baseline; 1, 3, 6, and 12 months postoperatively
  Upper extremity functional index-15 (UEFI-15) iss used to assess the functional status of the upper extremity by 15-items based on activities of daily living. Sum of the item scores are converted to final score between 0-100 points means the higher score is better functional capacity.
Exercise Adherence | Throughout the 12-month follow-up
  Compliance with the prescribed home-based exercise program is questioned if they are performing the exercises properly according to the template they are given at every visit with physician and overlooked if patient requires. Percentage of patients performing regular exercise will be interpreted after 12-months follow-up.

CONTACTS AND LOCATIONS:
Locations (1):
- UHS Balikesir Ataturk Health and Application Center, Balıkesir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Toohey K, Hunter M, McKinnon K, Casey T, Turner M, Taylor S, Paterson C. A systematic review of multimodal prehabilitation in breast cancer. Breast Cancer Res Treat. 2023 Jan;197(1):1-37. doi: 10.1007/s10549-022-06759-1. Epub 2022 Oct 21. PMID 36269525
- [Result] Del Bianco N, Borsati A, Toniolo L, Ciurnielli C, Belluomini L, Insolda J, Sposito M, Milella M, Schena F, Pilotto S, Avancini A. What is the role of physical exercise in the era of cancer prehabilitation? A systematic review. Crit Rev Oncol Hematol. 2024 Jun;198:104350. doi: 10.1016/j.critrevonc.2024.104350. Epub 2024 Apr 18. PMID 38642726